CLINICAL TRIAL: NCT02568618
Title: Patient and Provider Confidence and Satisfaction With the Clinical Use of CYP Genetic Variability Analysis to Guide Analgesic Treatment: A Randomized, Controlled Pilot Study Using the Pain Medication and Mental Health DNA InsightTM Test.
Brief Title: Patient and Provider Confidence and Satisfaction With the Clinical Use of CYP Genetic Variability
Acronym: Genomics
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor pulled funding related to enrollment pace.
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 409729
Record Dates: First submitted 2015-09-24; First posted 2015-10-06 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-04

CONDITIONS: Pain
Keywords: Military; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate (Other): Subjects will receive the results of the Pain Medication DNA Insight (TM) test at Visit 1.
  Interventions: Genetic: Pain Medication DNA Insight (TM) test
- Delayed (Other): Subjects will receive the results of the Pain Medication DNA Insight (TM) test at Visit 4. After 3 months of standard treatment.
  Interventions: Genetic: Pain Medication DNA Insight (TM) test

INTERVENTIONS:
Genetic: Pain Medication DNA Insight (TM) test — The DNA insight test uses saliva to test the metabolism of certain pain and mental health medications to determine if the subject is a poor metabolizer, intermediate metabolizer or ultrarapid metabolizer.

SUMMARY:
This study utilizes the Medication DNA Insight™ tests for pain and mental health medications. We are testing the pain and mental health medications commonly used in pain treatment. Subjects will give a sample of saliva that will be tested for the metabolism of the different medications. Consented providers will be given the results of the test and can determine whether to change the subject's medication regimen. Providers and subjects will be ask to complete surveys both pre and post visits. The purpose is to examine provider and patient satisfaction, confidence and certainty of using the test results.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, interventional pilot study analyzing both providers' and patients' perceptions and responses to the DNA Insight test. Twelve military health system primary care providers and 4 of each provider's patients will be enrolled in the study. (12 providers and 48 patients total) Each provider's patients will be randomized into delayed treatment (Group A) or immediate treatment (Group B) at a 1:1 ratio. All patients receive the Pain Medication and Mental Health DNA InsightTM test (intervention). Results for patients in Group A will be given to the provider with a 3 month delay. Those in the 3 month delay will serve as a comparison group for the period prior to receiving intervention. Results for patients in Group B will be given to the provider without delay, 2-3 weeks after saliva sample collection. The provider will use the results of the Pain Medication and Mental Health DNA InsightTM test to evaluate whether changes of medications are indicated based on the individual patient's genetic profile. A measure of the provider's certainty, confidence, satisfaction, perception of care and global impression of change will be assessed at baseline, prior to obtaining the test results, and after obtaining the test results, as outlined in the data collection section. Patients' pain related self-reported outcomes, certainty, confidence and satisfaction will be assessed at baseline, prior to obtaining the DNA InsightTM test results, and after receipt and implementation of the test results, as described in the data collection section of the protocol.

At the baseline visit (Visit 0) each enrolled patient will provide a saliva sample for the Pain Medication DNA InsightTM test that identifies genetic variation in CYP metabolism. The providers and patients will be recruited from any of the Womack Army Medical Center's Primary Care Medical Homes and family practice clinics.

ELIGIBILITY:
Inclusion Criteria:

* Military healthcare system beneficiary enrolled in the Womack Army Medical Center Health Care System
* Age 18 or older
* Patient of the enrolled provider for at least 3 months.
* Persisting pain for at least 3 months, with average daily pain score of 4 or higher that is not expected to improve without directed therapy.
* No history of chronic liver or kidney disease

Exclusion Criteria:

* Known pregnancy or breast feeding
* Planned deployment, permanent change of station, or military separation within upcoming 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Provider Satisfaction, Certainty and Confidence survey | 6 months
  Examine trends in provider decisions in prescribing analgesics and modifying analgesic treatment plans and provider outcomes for satisfaction, certainty and confidence in dosing of analgesics with and without access to Pain Medication and Mental Health DNA Insight ™ genetic testing results. A certainty, confidence, satisfaction survey, provider perception of care and provider global impression of change surveys will be administered to the provider after each visit from each study subject.
Provider perception of care survey | 6 months
  Examine trends in provider decisions in prescribing analgesics and modifying analgesic treatment plans and provider outcomes in perception of care
Provider global impression of change survey | 6 months
  Examine trends in provider decisions in prescribing analgesics and modifying analgesic treatment plans and provider outcomes for global impression of change

SECONDARY OUTCOMES:
Patient certainty, confidence and satisfaction survey | 6 months
  Examine trends in patients' satisfaction, certainty and confidence in dosing of analgesics between patient groups whose providers had access to Pain Medication and Mental Health DNA Insight ™ genetic testing results and those whose providers did not have access to the genetic information.
Patient perception of care survey | 6 months
  Examine trends in patient perception of care in dosing of analgesics between patient groups whose providers had access to Pain Medication and Mental Health DNA Insight ™ genetic testing results and those whose providers did not have access to the genetic information.
Patient global impression of change survey | 6 months
  Examine trends in patients' global impression of change in dosing of analgesics between patient groups whose providers had access to Pain Medication and Mental Health DNA Insight ™ genetic testing results and those whose providers did not have access to the genetic information.
Patient Outcomes pain as assessed by the DVPRS | 6 months
  Compare patient-reported pain between patient groups whose providers had early access to Pain Medication and Mental Health DNA Insight ™ genetic testing results to those who had delayed access in the control period and subsequently following later access to the results. Subjects will be ask to complete the DVPRS pain scale, a visual analog scale.
Patient Outcomes pain as assessed by BPI perception of pain relief item | 6 months
  Compare patient-reported pain between patient groups whose providers had early access to Pain Medication and Mental Health DNA Insight ™ genetic testing results to those who had delayed access in the control period and subsequently following later access to the results. Subjects will be ask to complete the BPI perception of pain relief item prior to each provider visit.
Patient Outcomes pain as assessed by the PROMIS Pain short form | 6 months
  Compare patient-reported pain between patient groups whose providers had early access to Pain Medication and Mental Health DNA Insight ™ genetic testing results to those who had delayed access in the control period and subsequently following later access to the results. Subjects will be ask to complete the PROMIS pain interference short forms prior to each provider visit.
Patient Outcomes of demographics | 6 months
  Compare patient-reported demographics for equality in sampling
Patient Outcomes of depression as assessed by the PROMIS depression short form | 6 months
  Compare patient-reported depression between patient groups whose providers had early access to Pain Medication and Mental Health DNA Insight ™ genetic testing results to those who had delayed access in the control period and subsequently following later access to the results. Subjects will be ask to complete the PROMIS depression short form prior to each provider visit.
Patient Outcomes of anxiety as assessed by the PROMIS anxiety short form | 6 months
  Compare patient-reported anxiety between patient groups whose providers had early access to Pain Medication and Mental Health DNA Insight ™ genetic testing results to those who had delayed access in the control period and subsequently following later access to the results. Subjects will be ask to complete the PROMIS anxiety short form prior to each provider visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bartoszek, MD, Principal Investigator — United States Department of Defense
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT02568618/Prot_SAP_000.pdf